CLINICAL TRIAL: NCT03878745
Title: Comparative User Experiences With BD Nano™ PRO 32G Extra Thin Wall Pen Needle vs the Terumo Nanopass® 34G Pen Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DBC-18PENDL01
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: BD Nano™PRO (Test Device) will be compared to the Terumo Nanopass® through a series of randomized abdominal saline injections
Masking Description: Participants will not see any labeling for the pen needles used for injections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BD Nano™ PRO 32G pen needle (Experimental): Participants are to perform 6 pairs of injections.
  Interventions: Device: Terumo Nanopass® 34G pen needle; Device: BD Nano™ PRO 32G pen needle
- Terumo Nanopass® 34G pen needle (Active Comparator): Participants are to perform 6 pairs of injections.
  Interventions: Device: Terumo Nanopass® 34G pen needle; Device: BD Nano™ PRO 32G pen needle

INTERVENTIONS:
Device: Terumo Nanopass® 34G pen needle — Insulin pen needle
Device: BD Nano™ PRO 32G pen needle — Insulin pen needle

SUMMARY:
This is a subject single blinded, block randomized, prospective, single-visit, multi-center study to compare user experiences with BD Nano™ PRO pen needle vs. the thinner commercially available Terumo Nanopass® pen needle. The study will include a minimum of 55 Japanese American study subjects with Type 1 or Type 2 diabetes.

DETAILED DESCRIPTION:
Study conduct will consist of one 60 to 120-minute Site visit in which pre-set doses of saline will be abdominally delivered by Subjects via a reusable insulin pen device. All pen needles will be attached by Study Staff and pen needle outer cover and inner shield will be removed for subjects. Subjects are to perform 12 injections into the abdomen (6 pairs of injections). Pairs of injections will be evaluated and each pair will contain one BD Nano™ PRO and one Terumo Nanopass® pen needle. The order of the two pen needles in each pair will be randomized.

The intent of this comparative use study is to determine whether Japanese American patients' experiences are different when using the BD Nano™ PRO 4mm x 32G extra thin wall, 5-bevel pen needle vs the Terumo Nanopass® 4mm x 34G pen needle in the Japanese American population. These experiences include the perceived force to deliver dose, the ability to deliver the full dose (measured by leakage), injection pain and bending.

ELIGIBILITY:
Inclusion Criteria:

1. Self-attesting Japanese American adults 18 to 75 years of age (inclusive).
2. Self-attest to Japanese descent.
3. Diagnosed with Type 1 or Type 2 diabetes.
4. Self-injecting using an injection pen for ≥3 months with any pen needle.
5. Injecting a minimum of ≥10 units of insulin and/or Victoza at least once per day.
6. Able to demonstrate proficiency using an injection pen into an injection model.
7. Able and willing to provide informed consent.
8. Able and willing to complete all study procedures.

Exclusion Criteria:

1. Not self-injecting (for example injections completed by a family member).
2. Self-injecting with a pen injector for less than 3 months.
3. Unwilling to inject into abdomen.
4. Unwilling to have hair at the injection area reduced with an electric razor if it is determined the hair will interfere with leakage evaluation.
5. Failure to confirm which pen needle (gauge and needle length) subject is currently using. To confirm, subject may be asked to bring their pen and pen needles to the site or site staff may confirm via medical record or pharmacy.
6. Pregnant (self-attestation).
7. Currently taking anti-platelet or anticoagulant therapy (up to 162 mg per day of aspirin is permitted).
8. History of a bleeding disorder.
9. History of recurrent dermatological conditions or skin disorder (e.g., psoriasis, eczema).
10. Gross skin anomalies and abnormalities located at or very close to the injection sites that would significantly limit available injection space.
11. History of symptomatic low blood pressure or history of fainting (syncope) during hypodermic injections.
12. Use of any analgesic medications within 24 hours of first study injection, and during the study (up to 162 mg per day of aspirin is permitted).
13. A current or previous medical or physical condition that, in the opinion of the investigator, would place the patient at risk or make them unable to perform study procedures or has the potential to confound interpretation of the study results.
14. Currently participating in another pen needle study.
15. Employed by, or currently serving as a contractor or consultant to BD or any diabetes injectable medication, injection pen, or pen needle manufacturer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mills-Peninsula Medical Center Dorothy L. and James E Frank Diabetes Research Institute, San Mateo, California
  - East West Medical Research Institute, Honolulu, Hawaii

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edwards CL, Fillingim RB, Keefe F. Race, ethnicity and pain. Pain. 2001 Nov;94(2):133-137. doi: 10.1016/S0304-3959(01)00408-0. PMID 11690726
- [Background] Watson PJ, Latif RK, Rowbotham DJ. Ethnic differences in thermal pain responses: a comparison of South Asian and White British healthy males. Pain. 2005 Nov;118(1-2):194-200. doi: 10.1016/j.pain.2005.08.010. Epub 2005 Oct 3. PMID 16202529
- [Background] Palmer B, Macfarlane G, Afzal C, Esmail A, Silman A, Lunt M. Acculturation and the prevalence of pain amongst South Asian minority ethnic groups in the UK. Rheumatology (Oxford). 2007 Jun;46(6):1009-14. doi: 10.1093/rheumatology/kem037. Epub 2007 Mar 31. PMID 17401133
- [Background] Komiyama O, Kawara M, De Laat A. Ethnic differences regarding tactile and pain thresholds in the trigeminal region. J Pain. 2007 Apr;8(4):363-9. doi: 10.1016/j.jpain.2006.12.002. Epub 2007 Feb 1. PMID 17275416
- [Background] Hobara M. Beliefs about appropriate pain behavior: cross-cultural and sex differences between Japanese and Euro-Americans. Eur J Pain. 2005 Aug;9(4):389-93. doi: 10.1016/j.ejpain.2004.09.006. PMID 15979019
- [Derived] Gibney MA, Fitz-Patrick D, Klonoff DC, Whooley S, Lu B, Yue W, Glezer S. User experiences with second-generation 32-gauge x 4 mm vs. thinner comparator pen needles: prospective randomized trial. Curr Med Res Opin. 2020 Oct;36(10):1591-1600. doi: 10.1080/03007995.2020.1803248. Epub 2020 Aug 18. PMID 32723109

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Subjects are to perform 6 pairs of injections. Each Pair consists of BD Nano™ PRO pen needle vs Terumo
Period: Overall Study
Arm/Group | All Study Participants
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 55
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Are you of Japanese descent [Count of Participants; unit: Participants]
  Yes | 55
  No | 0
Born in Japan [Count of Participants; unit: Participants]
  Yes | 9
  No | 46
At Least one(1) Parent born in Japan [Count of Participants; unit: Participants]
  Yes | 12
  No | 43
At Least one(1) Grandparent born in Japan [Count of Participants; unit: Participants]
  Yes | 51
  No | 4

OUTCOME MEASURES:

1. Primary Outcome: BD Nano™ PRO Pen Needle Compared to Terumo Nanopass® (Injection Pain)
Description: Injection pain as measured by a relative 150mm visual analog scale. Injection pain as measured by a relative visual analog scale. s. User preference is assessed through a single question reported on a 150mm relative VAS scale with the BD Nano™ PRO pen needle Pen labeled at +75 mm and the Comparator pen needle labeled at -75mm. On this scale, zero represents no preference to either pen needle. Relative VAS scores range from -75mm to 75mm; positive scores reflect preference forBD Nano™ PRO and negative scores reflect preference for the comparator.
  Scores from each of the paired injections (330 pairs for all participants) were pooled and a mean was calculated. The two-sided 95% confidence interval was calcuated for the average relative rating. A linear model was used to adjust for the order effect.
  If the lower bound of the 95% CI is > -10cm, non-inferiority could be concluded. If the lower bound of the 95% CI is >0, superiority can also be concluded.
Time Frame: Scores were collected immediately after each paired injection
Population: Per protocol population
Measure: Mean (95% Confidence Interval); unit: mm
Units Other Than Participants: paired injections
Arm/Group | All Study Participants
Number analyzed (Participants) | 55
Number analyzed (paired injections) | 330
mm | 7.30 [2.2 to 12.39]

2. Secondary Outcome: BD Nano™ PRO vs Terumo Nanopass® (Force)
Description: Subject perceived force required to deliver dose measured by a relative 5 point Likert scale. The scale ranged from -2 to 2, where positive scores indicated less thumb force required for the BD Nano™ PRO, and negative scores indicated less thumb force for Terumo Nanopass®. Scores from each of the paired injections (330 pairs for all participants) were pooled and a mean was calculated.
Time Frame: Scores were collected immediately after each paired injection
Population: Per-protocol population
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: paired injections
Arm/Group | All Study Participants
Number analyzed (Participants) | 55
Number analyzed (paired injections) | 330
score on a scale | 0.210 [0.07 to 0.35]
Statistical Analysis 1: Comparison: All Study Participants; Test type: Superiority — Two-sided 95% confidence intervals is calculated for the average relative rating. A linear model was used to evaluate the pen needle group effect on the response to test whether the groups can be combined and to adjust for the order effect. The order of the pen needles used and the group to which the subject belongs were used as covariates. If the lower bound of the CI is > 0, we can conclude in superiority; Overall Mean = 0.210, 95% CI 2-sided [0.07 to 0.35]

3. Secondary Outcome: BD Nano™ PRO vs Terumo Nanopass® (Needle Bending)
Description: Participants reported a visual score of needle bending. A score of at least 2, corresponding to >10 degrees of bending, was considered an event of a bent needle. The percentage of of bending events (yes/no) was calculated for each groups and the mean difference calculated along with a 95% confidence interval.
Time Frame: Immediately after injections were completed
Population: per protocol population
Measure: Number (95% Confidence Interval); unit: percentage of needles with bending
Units Other Than Participants: pen needles
Groups:
- BD Nano™ PRO; Terumo Nanopass: All participants received 6 paired injections.
Arm/Group | BD Nano™ PRO | Terumo Nanopass
Number analyzed (Participants) | 55 | 55
Number analyzed (pen needles) | 330 | 330
percentage of needles with bending | 0.6 [0.2 to 2.5] | 0.6 [0.2 to 2.2]
Statistical Analysis 1: Comparison: BD Nano™ PRO vs Terumo Nanopass; Test type: Other; Mean Difference (Final Values) = 0, 95% CI 2-sided [-1.6 to 1.6]

4. Secondary Outcome: BD Nano™ PRO vs Terumo Nanopass® (Leakage)
Description: After saline delivery equivalent to 30U of U100 insulin (0.3mL) and subject removal of pen needle from body, study staff used the provided materials and scale to absorb leakage from the pen needle tip and injection site to measure the amount of leakage. Leakage over 0.015g was counted as an event. The percentage of of leakage events (yes/no) was calculated for each groups and the mean difference calculated along with a 95% confidence interval.
Time Frame: Immediately after injection
Population: per protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants with leakage
Units Other Than Participants: Pen Needles
Groups:
- BD Nano™ PRO; Terumo Nanopass: Subjects are to perform 6 pairs of injections. Each Pair consists of BD Nano™ PRO pen needle vs Terumo
Arm/Group | BD Nano™ PRO | Terumo Nanopass
Number analyzed (Participants) | 55 | 55
Number analyzed (Pen Needles) | 330 | 330
percentage of participants with leakage | 0.3 [0 to 1.7] | 1.8 [0.8 to 3.9]
Statistical Analysis 1: Comparison: BD Nano™ PRO vs Terumo Nanopass; Test type: Other; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-3.6 to 0.1]

5. Other Pre Specified Outcome: Compare BD Nano™ PRO vs Terumo Nanopass® (Total Injection Time)
Description: Time from when injection button fully depressed to when pen needle removed from body. Mean total injection time was calculated for both the BD Nano™ PRO and the Terumo Nanopass®. Scores from each injection (330 for each needle type) were pooled and a mean was calculated. The total injection time for the BD Nano™ PRO and Terumo Nanopass® were compared and the mean difference reported with a 95% confidence interval.
Time Frame: Immediately after injections were completed
Population: Per Protocol population
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: pen needles
Arm/Group | All Study Participants
Number analyzed (Participants) | 55
Number analyzed (pen needles) | 660
seconds
  BD NANO: number analyzed (pen needles) | 330
  BD NANO | 7.55 (4.75)
  Terumo: number analyzed (pen needles) | 330
  Terumo | 7.80 (4.62)
Statistical Analysis 1: Comparison: All Study Participants; Test type: Superiority — A mixed effect model was used (fixed effects of PN, abdomen site, order of pair, order of PN within pair and random subject effect) to estimate average difference (BD Nano PN - Terumo PN) in delivery time and total injection time. A Box-Cox transformation might be used to normalize the data if necessary; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -0.50, 95% CI 1-sided [upper limit -0.026]

6. Other Pre Specified Outcome: Compare BD Nano™ PRO vs Terumo Nanopass® (Needle Breaking)
Description: Needle breakage was defined as the patient-end metal cannula being separated into two pieces. The percentage of of breaking events (yes/no) was calculated for each groups and the mean difference calculated along with a 95% confidence interval.
Time Frame: Immediately after injections were completed
Population: Per-protocol population
Measure: Number (95% Confidence Interval); unit: percentage of needles with breaking
Units Other Than Participants: pen needles
Groups:
- BD Nano™ PRO: Subjects are to perform 6 pairs of injections.
- Terumo Nanopass: All participants are to perform 6 pairs of injections
Arm/Group | BD Nano™ PRO | Terumo Nanopass
Number analyzed (Participants) | 55 | 55
Number analyzed (pen needles) | 330 | 330
percentage of needles with breaking | 0 [0 to 1.1] | 0 [0 to 1.1]
Statistical Analysis 1: Comparison: BD Nano™ PRO vs Terumo Nanopass; Test type: Other; Mean Difference (Final Values) = 0, 95% CI 2-sided [-1.2 to 1.2]

7. Post Hoc Outcome: Subject Satisfaction Survey
Description: Each subject was asked to fill out a 4 question survey on the general importance of Injection Pain, Thumb pressure, Leakage and Needle Bending, each question was tabulated. Each participant answered 1 survey about their general preferences and opinions, not regarding either product used in the study.
Time Frame: Immediately after injections were completed
Population: Each subject was asked to fill out a 4 question survey on the importance of Injection Pain, Thumb pressure, Leakage and Needle Bending
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: Subject Satisfaction Survey
Arm/Group | All Study Participants
Number analyzed (Participants) | 55
Participants
  Injection Pain affects my level of satisfaction: Agree | 16
  Injection Pain affects my level of satisfaction: Somewhat Agree | 16
  Injection Pain affects my level of satisfaction: Neutral | 16
  Injection Pain affects my level of satisfaction: Somewhat Disagree | 3
  Injection Pain affects my level of satisfaction: Disagree | 4
  Thumb pressure needed affects my level of satisfac: Agree | 10
  Thumb pressure needed affects my level of satisfac: Somewhat Agree | 21
  Thumb pressure needed affects my level of satisfac: Neutral | 14
  Thumb pressure needed affects my level of satisfac: Somewhat Disagree | 7
  Thumb pressure needed affects my level of satisfac: Disagree | 3
  Post injection leakage increases level of concern: Agree | 18
  Post injection leakage increases level of concern: Somewhat Agree | 16
  Post injection leakage increases level of concern: Neutral | 16
  Post injection leakage increases level of concern: Somewhat Disagree | 4
  Post injection leakage increases level of concern: Disagree | 1
  A bent needle increases my level of concern: Agree | 23
  A bent needle increases my level of concern: Somewhat Agree | 13
  A bent needle increases my level of concern: Neutral | 17
  A bent needle increases my level of concern: Somewhat Disagree | 1
  A bent needle increases my level of concern: Disagree | 1

ADVERSE EVENTS:
Time Frame: For each subject, adverse event data was collected at one visit.
Groups:
- Terumo Nanopass: Subjects are to perform 6 pairs of injections.
Arm/Group | BD Nano™ PRO | Terumo Nanopass
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT03878745/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT03878745/SAP_001.pdf